CLINICAL TRIAL: NCT07085585
Title: The Embryo-endometrium Multifaceted Interface: Endometrial Cavity Molecular Microbiobial and Transcriptomic Signatures in Predictinf Pregnancy Outcome in Infertile Patients Undergoing Assisted Reproduction Technology Procedures
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Rovere Querini Patrizia, MD, PhD, IRCCS San Raffaele
Other Study IDs: RF-2019-12369460; RF-2019-12369460 (Other Grant/Funding Number: Ministry of Health (Italy))
Record Dates: First submitted 2025-06-13; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Infertility (IVF Patients)
Keywords: Extracellular Vesicles; endometrial microbiome; RNA-Seq
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Uterine fluid samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fertile women: Reference group
- infertile women undergoing ART cycles: Cases group

SUMMARY:
In reproductive medicine, a fundamental challenge is to evaluate the endometrial health status during the embryo implantation window as a limiting step in predicting the success of treatments of assisted reproduction technology (ART). Some highthroughput tools, recently developed by private genomics companies, are available in the market even if they have not been independently validated and have different limitations. We propose a prospective cohort study with the aim of validating the reliability and increasing efficacy of these tools. Endometrial fluid samples will be collected non-invasively from women undergoing ART cycles and isolated genetic materials will be subjected to 16S rRNA gene sequencing for microbiota profiling and to RNAseq analysis of RNA content of extracellular vesicles previously recognized as a tissue proxy in predicting endometrial receptivity. Clinical pregnancy rate/first cycle will be the target outcome used to assess the resulting predictive models. Ultrasonographic features of the endometrium will also be collected and accounted for in the predictive model.

ELIGIBILITY:
IVF Patients inclusion Criteria:

* Indication to ART
* Age 18-39 years
* First ART cycle
* Normal uterine morphology and no hydrosalpinx at ultrasound

IVF Patients exclusion Criteria:

* Poor responders according to Bologna criteria
* Indications to ART for severe male infertility

Fertile Patients inclusion Criteria:

* Subjects will be cycling women with proven fertility undergoing laparoscopy for tubal ligation
* BMI < 30
* Aged 20 to 40 years

Fertile Patients exclusion Criteria:

* Smokers
* Not taking any medication

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study population is composed of women undergoing assisted reproduction treatments, specifically in vitro fertilization (IVF). These patients are followed in an outpatient setting at two specialized infertility centers in Italy: San Raffaele Hospital and Fondazione Cà Granda Policlinico. They are women who have been referred to IVF due to infertility, and are starting their first IVF cycle. All participants meet specific inclusion criteria, such as being between 18 and 39 years of age, having normal uterine anatomy, and no evidence of hydrosalpinx on ultrasound examination.
  The outpatient nature of the study allows for non-invasive sampling procedures and routine follow-up without the need for hospitalization. This setting reflects real-world clinical practice in reproductive medicine, ensuring that the findings will be directly applicable to standard IVF care. Additionally, the study includes a group of fertile women, also managed on an outpatient basis, who serve as a reference.
Sampling Method: Non-Probability Sample
Enrollment: 322 (Estimated)
Dates: Start 2021-01-24 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Identification of endometrial microbiome diversity | through study completion, an average of 1 year
  Evaluation of the endometrial microbiome composition and diversity using 16S rRNA sequencing to assess the functional impact of the endometrial microbial community in predicting the clinical pregnancy rate in women undergoing ART cycles.
Extracellular Vesicle (EV) RNA Profiles | through study completion, an average of 1 year
  Quantification of extracellular vesicle (EV) RNA expression profiles from uterine fluid samples using RNA sequencing (expressed in CPM). Confirmation of the good correlation between expression of genes in tissue samples and in endometrial-derived EVs.
Integrated Predictive Model for Clinical Pregnancy | through study completion, an average of 1 year
  Development of a multivariable predictive model combining endometrial microbiome diversity, EV RNA profiles, and ultrasound-AI analysis to predict clinical pregnancy rates in ART cycles.

CONTACTS AND LOCATIONS:
Locations (1):
- OSR Innate Immunity and tissue remodeling Unit and Centro Scienze Natalità OS, Milan, milano, Italy

IPD SHARING:
Plan to Share IPD: No